CLINICAL TRIAL: NCT06680323
Title: Identification of Risk Factors, Exposomics and Genetic Susceptibility of Melanoma in Children, Adolescents and Young Adults - Novel Health Care Strategies for Melanoma in Children, Adolescents and Young Adults (MELCAYA)
Brief Title: Identification of Risk Factors, Exposomics and Genetic Susceptibility of Melanoma in Children, Adolescents and Young Adults
Acronym: ExpoMel
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Hospital Clinic of Barcelona (Other); University Of Perugia (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Karolinska University Hospital (Other); Leibniz Research Institute for Environmental Medicine Düsseldorf (Unknown); Princess Maxima Center for Pediatric Oncology (Other); Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: 834/2023BO2
Record Dates: First submitted 2024-09-25; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-09

CONDITIONS: Melanoma; Spitzoid Melanoma; Congenital Nevi
Keywords: etiology; melanoma; children; adolescents; young adults; genetic predisposition; epidemiology; exposomes
MeSH Terms: conditions — Melanoma; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue samples of melanoma and normal tissue, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Classic melanoma: Classic malignant melanoma under the age of 30 years For patients with available biospecimen, the germline genome, transcriptome and in selected cases tumour normal exomes will be sequenced.
- Spitzoid melanoma: Spitzoid melanoma under the age of 30 years For patients with available biospecimen, the germline genome, transcriptome and in selected cases tumour normal exomes will be sequenced.
- Other melanoma: Other melanoma as melanoma on congenital nevi under the age of 30 years For patients with available biospecimen, the germline genome, transcriptome and in selected cases tumour normal exomes will be sequenced.

SUMMARY:
The primary objective of this study is the identification of environmental and genetic factors involved in the risk and progression of melanoma in children, adolescents and young adults (CAYA). The secondary objectives are to generate a model integrating the genetic and environmental factors to estimate the risk of developing melanoma and improve the primary prevention of melanoma through evidence-based interpretation of environmental risk.

DETAILED DESCRIPTION:
By retrieving data from several epidemiological and clinical registries across Europe it is aimed to integrate and maximize efforts in order to create a large dataset that serves for a comprehensive analysis of genetic and environmental factors influencing the etiology of melanoma in CAYA. The data will be combined with exposome information about climate and pollution for the development of a weighted risk score. Furthermore, germline high risk mutations and germline low-medium risk variants will be analyzed. Genome and transcriptome sequencing of blood and in selected cases tumour will provide the most comprehensive data to create a polygenic risk score for CAYA melanoma. Transcriptome data will help to identify and characterize the effect of variants of unknown significance in coding, intronic as well as regulatory regions. Tumour sequencing can provide additional information on functional relevance of variants, e.g. secondary hits in tumour tissue or second hits in tumour suppressor genes. Such identification will be highly advantageous to design prevention strategies for melanoma development in CAYA.

ELIGIBILITY:
Inclusion Criteria:

* confirmed melanoma
* age until 30 years old

Exclusion Criteria:

* no available biological material
* no signed informed consent

Max Age: 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: Due to its registry-based retrospective study, no formal recruitment of patients will occur in ExpoMel. Data and samples will be obtained from the following registries and associated biobanks:
  * Catalonia Melanoma Network through Hospital Clinic Barcelona
  * The German Registry for Rare Pediatric Tumours (STEP) of the German Society for Pediatric Oncology and Hematology
  * Swedish Melanoma Registry (SweMR) through Karolinska Institute
  * Public Pathology Database of the Netherlands (PALGA) through Princess Maxima Center for Children OncologyCentral Registry Malignant Melanoma of the German Dermatological Society (CMMR)
  * Polish Pediatric Rare Tumor Study group and selected Eastern/Southern Europe countries cooperating within the European Cooperative Study Group for Pediatric Rare Tumors (EXPERT) through the Medical University Gdansk
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Identification of environmental and genetic factors involved in the risk and progression of melanoma in children, adolescents and young adults (CAYA) | 01.01.2024 - 30.11.2025
  By retrieving data from several epidemiological and clinical registries across Europe we aim to create a large dataset that serves for a comprehensive analysis of genetic and environmental factors influencing the etiology of melanoma in CAYA. Data on climate variables such as surface temperature, solar radiation, and air pollutants will be collected from ground-based instruments, such as air quality monitoring stations, and satellites and reanalysis data from the Copernicus Atmosphere Monitoring Service (CAMS). Data analysis from genome sequencing will be done using established bioinformatic pipelines and combined with exposome information about climate and pollution for the development of a weighted risk score.

SECONDARY OUTCOMES:
Generating a polygenic risk score for melanoma in CAYA by using the Lindeman-Merenda-Gold (LMG) method | 01.06.2024 - 31.05.2026
  Genome and transcriptome sequencing of blood and in selected cases tumour will provide the most comprehensive data to create a polygenic risk score for melanoma in CAYA.
  We will develop a weighted risk score for each environmental factor, which comprises the effects of several variables measuring the respective risk factor. Additionally, a weighted risk score for the epigenetic variables will be build. To estimate the relative contribution of environmental and epigenetic factors we will calculate the relative importance (proportion of explained variance) of the weighted risk scores in an ordinary linear regression model using the Lindeman-Merenda-Gold (LMG) method.
Prevention strategies for melanoma development in CAYA | 01.06.2025 - 30.09.2026
  The detected risk factors and determinants will be used by health professionals to update clinical guidelines for prevention, screening and early detection of melanoma in CAYA. Health care system strategies will be implemented in European countries overcoming current gaps in European countries on prevention and diagnosis of melanoma in CAYA. The success will be measured by incidence rates of melanoma.

CONTACTS AND LOCATIONS:
Locations (6):
- Leibniz Research Institute for Environmental Medicine, Düsseldorf, Germany
- Italy (2):
  - University of Florence, Florence
  - Istituto Nazionale del Tumori, Milan
- Medical University of Gdánsk, Gdansk, Poland
- Hospital Clínic de Barcelona, Barcelona, Spain
- Karolinska Institute, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Undecided